CLINICAL TRIAL: NCT04860063
Title: Effect of Berberine on Metabolic Syndrome, Efficacy and Safety in Combination With Antiretroviral Therapy in People Living With HIV.
Brief Title: Effect of Berberine on Metabolic Syndrome, Efficacy and Safety in Combination With Antiretroviral Therapy in PLWH.
Acronym: BERMESyH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Shaúl Ariel Navarro Lara, Resident, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MeSHIV-001
Record Dates: First submitted 2021-04-17; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Metabolic Syndrome; HIV-1-infection; Glucose Intolerance; Dyslipidemias; Lipodystrophy; Lipoatrophy
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance; Dyslipidemias; Lipodystrophy | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo three times daily for 6 months
  Interventions: Drug: Placebo
- Berberine (Experimental): Berberine 500 mg three times daily for 6 months
  Interventions: Drug: Berberine

INTERVENTIONS:
Drug: Berberine — Participants randomly assigned to the intervention group will be provided with Berberine 500 mg administrated per os three times a day for six months
  Arms: Berberine
Drug: Placebo — Participants randomly assigned to the Placebo group will be provided with placebo administrated per os three times a day for six months
  Arms: Placebo

SUMMARY:
With current antiretroviral therapy, people living with HIV reach virological suppression faster, which in turn leads to a higher life expectancy. Nevertheless, this improved survival rate is not free of other comorbidities, such as metabolic syndrome, characterized by a decrease in glucose tolerance and an increase in insulin resistance.

Berberine is an alkaloid that has proven beneficial effects on both glucose tolerance and insulin resistance, but has not been tested in people living with HIV under virological suppression. We hypothesize that berberine will improve inflammatory markers and metabolic profile in this population without significant interactions nor adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Documented HIV-1 infection
* Stable antiretroviral therapy at least 6 months before enrollment
* Viral suppression
* Metabolic syndrome , defined by Adult Treatment Panel-III criteria
* No previously known kidney or liver disease
* Signed informed consent

Exclusion Criteria:

* People younger than 18 years and older than 60 years
* Prior atherosclerotic cardiovascular disease
* Diabetes mellitus type 1 or 2
* Previous use of glucose and/or lipid modifying medications
* Pregnancy
* Withdrawal of informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | 24 weeks within randomization
  Change from Baseline insulin resistance determined by Homeostasis Model Assessment index, triglyceride to glucose ratio, at 6 months
Change from baseline lipid profile at 6 months | At the beginning and 24 weeks within randomization
  Measurement of total cholesterol, HDL, LDL, triglycerides.

SECONDARY OUTCOMES:
Change from baseline weight | At the beginning and 24 weeks within randomization
  Weight gain or loss measure by kilograms
Inflammatory profile | At the beginning and 24 weeks within randomization
  Level of pro-inflammatory cytokines

REFERENCES:
- [Derived] Ruiz-Herrera VV, Navarro-Lara SA, Andrade-Villanueva JF, Alvarez-Zavala M, Sanchez-Reyes K, Toscano-Pina M, Mendez-Clemente AS, Martinez-Ayala P, Valle-Rodriguez A, Gonzalez-Hernandez LA. Pilot study on the efficacy and safety of berberine in people with metabolic syndrome and human immunodeficiency virus infection. Int J STD AIDS. 2023 Dec;34(14):1042-1052. doi: 10.1177/09564624231196600. Epub 2023 Aug 23. PMID 37611246